CLINICAL TRIAL: NCT06016140
Title: Applying a Medication Plan for Safer Medication Treatment in Older Persons - a Feasibility Study
Brief Title: A Medication Plan for Safer Medication Treatment in Older Persons
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Jönköping County (Other Government)
Collaborators: Jonkoping University (Other)
Responsible Party: Principal Investigator, Malin Holmqvist, PhD student, pharmacist, Region Jönköping County
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022-04430-01
Record Dates: First submitted 2023-06-20; First posted 2023-08-29 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Patient Safety
Keywords: aged; medication; feasibility study; primary care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Medication Plan Prototype
  Interventions: Other: Medication plan

INTERVENTIONS:
Other: Medication plan — Involved participants will jointly agreed on continued medication treatment (treatment aim, planned monitring and evaluation and responsibility, and the physician will document the plan in the electronic health record

SUMMARY:
Harm from medications is still a concern in an aged population. As medication treatment for older persons many times are complex, a feasibility study can be helpful to support decisions about future evaluation and implementation of an intervention.

In this study, the overall aim is to assess feasibility, acceptability and potential effects of usage of a co-designed medication plan for older persons with medication treatment.

The study will take place in the primary care setting in Sweden, and involve persons 75 years or older using five or more medications on daily basis, physicians at primary care centers and persons supporting the older person in their medication use a home.

During an appointment, the physician and older person will agree on a medication plan, that will be documented in the older person's electronic health record and printed out on paper.

After three month, the potential outcomes of a medication plan will be collected, together with data about feasibility and acceptability of the intervention. Two questionnaires will be used, addressing usability and patient safety. Moreover, remote interviews with participants will be performed to address usability and patient safety. Information about the medication plan will be collected from the electronic health record. Data analysis will be done with descriptive statistics and qualitative content analysis.

Expected outcomes are an assessment of feasibility and acceptability, and potential outcomes, to support decision on a future evaluation of the medication plan.

ELIGIBILITY:
Inclusion Criteria:

* Physicians and nurses: regular contact with the older person regarding medications, employment at a primary care center and ability to understand and communicate in Swedish
* Older persons: age >75 years old, five or more medications on a regular basis and ability to understand and communicate in Swedish
* Next-of-kin: age > 18 years old, regular contact with the older person regarding medications, ability to understand and communicate in Swedish

Exclusion Criteria:

* Older persons: impaired cognitive ability affecting the ability to provide informed consent (Diagnosis code for dementia) and late palliative phase, here defined as estimated life expectancy shorter than six months
* Next-of-kin: impaired cognitive ability affecting the ability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of the intervention | Three months
  For feasibility of the intervention, the secondary outcome measures will be analyzed together to address the feasibility of chosen study methods and of the intervention of using a co-designed medication plan

SECONDARY OUTCOMES:
Usability of the medication plan | Three months
  A modified version of Brookes "The System Usability Scale, SUS" will be used to measure usability of the medication plan. SUS is a widely used questionnaire for measuring the perception of the user experience and has been translated and evaluated in Swedish. The questions will be distributed by e-mail or mail (which is preferred of the participants) at the end of the three-month follow-up period.
Usability of the medication plan | Three months
  Semi-structured interviews, with questions addressing usability will be conducted with participants (older persons, next-of-kin, physicians, nurses) at the end of the three-month follow-up period. The interview guide will be guided by topics addressed in SUS. A strategic selection of all participants will be used to gather different experiences. The interviews will be audio-recorded and then will be transcribed verbatim.
Patient safety | Three months
  We will use a selected number of questions, which addresses concerns related to safety, from the Swedish National Patient survey in primary care, and ask the older persons to complete the questionnaire. No similar measurement will be used for healthcare professionals and next-of-kin.
Patient safety | Three months
  We will complement the questionnaire with semi-structured interviews performed with older persons, nurses, next-of-kin and physicians. Questions addressing patient safety will be asked to the same population and at the same occasion as the interviews about usability. The interview guide will be guided by questions in the Swedish National Patient survey and inspired by indicators for safety monitoring in healthcare as proposed by Vincent et al.
Acceptability of the intervention | Three months
  Acceptability of the intervention will be assessed by collecting the number of completed and adjusted medication plans, the content in the medication plans and medications prescribed for each older person during the follow up period
Healthcare utilisation | Three months
  Healthcare utilisation will be measured as number and cause, of hospital admission, emergency visits and unplanned physician visits during the follow up period

CONTACTS AND LOCATIONS:
Overall Officials: Malin Holmqvist, Principal Investigator — Region Jönköping County
Locations (1):
- Region Jonkoping County, Jönköping, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holmqvist M, Ros A, Thor J, Johansson L. Applying a co-designed medication plan for safer medication treatment in older persons: a feasibility study. Pilot Feasibility Stud. 2025 Jul 3;11(1):92. doi: 10.1186/s40814-025-01661-1. PMID 40611301